CLINICAL TRIAL: NCT02863614
Title: Analgesia for Endometrial Scratching in Subfertile Women: a Randomized Controlled Trial
Brief Title: Analgesia for Endometrial Scratching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Wellington P Martins, MD, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CAAE: 36622214.5.0000.5440
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Subfertility; Infertility
MeSH Terms: conditions — Infertility | interventions — Ibuprofen; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ibuprofen+Lorazepam (Experimental): Oral ibuprofen (600 mg) + lorazepam (1 mg); one hour before endometrial scratching.
  Interventions: Drug: Ibuprofen 600 mg; Drug: Lorazepam 1 mg
- Ibuprofen (Active Comparator): Oral ibuprofen (600 mg) + Placebo; one hour before endometrial scratching.
  Interventions: Drug: Ibuprofen 600 mg; Drug: Placebo
- Placebo (Placebo Comparator): Placebo + Placebo; one hour before endometrial scratching.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen 600 mg
  Arms: Ibuprofen; Ibuprofen+Lorazepam
Drug: Lorazepam 1 mg
  Arms: Ibuprofen+Lorazepam
Drug: Placebo
  Arms: Ibuprofen; Placebo

SUMMARY:
The aim of this study is to evaluate whether Ibuprofen alone or combined with lorazepam reduce the pain associated with endometrial scratching/injury.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years undergoing assisted reproduction (IUI, IVF/ICSI, frozen embryo transfer)
* Being submitted to endometrial scratching/injury with a Pipelle on the first four days of the menstrual cycle.
* Not have performed endometrial scratching in the last 90 days.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Maximum pain during procedure | 5 minutes
  Evaluated by both visual analog scale (10 cm) and numeric verbal scale (0 to 10).

SECONDARY OUTCOMES:
Pain after the procedure | 5 minutes
  Evaluated by both visual analog scale (10 cm) and numeric verbal scale (0 to 10).
Rejection to a new procedure | 5 minutes
  Evaluated by a 5-point Likert scale, commenting on this sentence: "I would repeat this procedure if it were indicated". 1 = I fully agree; 2 = I agree; 3 =Neither agree nor disagree; 4 = Disagree; 5 = Strongly Disagree.